CLINICAL TRIAL: NCT05967897
Title: Enhancing the Benefits of Blueberry Polyphenols With Plant and Whey Proteins
Brief Title: Enhancing the Benefits of Blueberry Polyphenols With Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 3647
Record Dates: First submitted 2023-06-22; First posted 2023-08-01 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Healthy Adults
Keywords: Healthy; Adults; Blueberries; Polyphenols; Protein; Bioavailability
MeSH Terms: interventions — blueberry extract; Whey Proteins; Pea Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blueberries (Experimental): Freeze-dried blueberry powder
  Interventions: Dietary Supplement: Blueberries
- Blueberries and Whey Protein (Active Comparator): Freeze-dried blueberry powder and whey protein
  Interventions: Dietary Supplement: Blueberries and Whey Protein
- Blueberries and Pea Protein (Active Comparator): Freeze-dried blueberry powder and pea protein
  Interventions: Dietary Supplement: Blueberries and Pea Protein
- Blueberries and Hemp Protein (Active Comparator): Freeze-dried blueberry powder and hemp protein
  Interventions: Dietary Supplement: Blueberries and Hemp Protein

INTERVENTIONS:
Dietary Supplement: Blueberries — 22 g freeze-dried blueberry powder mixed with water
  Arms: Blueberries
Dietary Supplement: Blueberries and Whey Protein — 22 g freeze-dried blueberry powder mixed with whey protein and water
  Arms: Blueberries and Whey Protein
Dietary Supplement: Blueberries and Pea Protein — 22 g freeze-dried blueberry powder mixed with pea protein and water
  Arms: Blueberries and Pea Protein
Dietary Supplement: Blueberries and Hemp Protein — 22 g freeze-dried blueberry powder mixed with hemp protein and water
  Arms: Blueberries and Hemp Protein

SUMMARY:
The purpose of this randomized crossover trial is determine whether acute consumption of blueberries with different proteins from plants (hemp or pea) or dairy (whey) impact the absorption of blueberry phytochemicals, which could impact the health benefits of blueberries. A secondary purpose is to understand the role that the gut microbiome may play, as well as the impact on urine polyphenol metabolites and potential implications for cardiometabolic health. Researchers will compare four arms: 1) Blueberries; 2) Blueberries + whey protein; 3) Blueberries + pea protein; and 4) Blueberries + hemp protein.

DETAILED DESCRIPTION:
Polyphenols are a structurally diverse class of secondary metabolites found in plants, with numerous documented benefits for human health including, but not limited to, anti-inflammatory, antioxidative and cardiovascular-protective effects. Dietary intake of polyphenols in the United States is low in comparison to other developed countries due to low intake of fruits and vegetables. Recent studies suggest fruit and vegetable intake should be increased by incorporating those foods into snacks and mixed meals as ingredients rather than standalone food items. Presently, berries comprise 10% of the total fruit intake and 7% of the total polyphenol intake of American adults. As a versatile food ingredient, berries can easily be added to foods like smoothies and yogurts as an ingredient to increase intake.

Low polyphenol intake is an issue exacerbated by poor bioavailability. Consumption does not necessarily mean that these beneficial compounds are delivered to body tissues, as evidenced by low levels of detection in blood and accumulation in the lower gastrointestinal tract after feeding. Bioavailability can be enhanced through the complexation of polyphenols with proteins, a phenomenon which occurs naturally in complex mixtures including both classes of nutrients. It has been shown that the complexation of polyphenols with proteins in cow's milk, known as a "matrix effect", enhances the polyphenol stability and uptake throughout digestion. The incorporation of berries into complex food mixtures may not only be an opportunity for improved health outcomes due to increased polyphenol intake, but also an effective strategy for ensuring that consumers receive the benefits of the nutrients they consume.

It is unknown whether the beneficial matrix effects observed when polyphenols interact with dairy proteins are exclusive to dairy proteins due to characteristics of high digestibility or structures which favor phenolic interaction, or if similar effects would be observed with proteins from other sources. Increasing consumer demand for alternative protein sources for reasons pertaining to human health and environmental sustainability has introduced a variety of novel plant-based proteins to the American diet, which may elicit similarly advantageous matrix effects on the bioavailability of polyphenols depending on their digestibility and structural characteristics. Understanding protein-polyphenol interactions in novel food matrices is necessary for the development of food products that promote polyphenol consumption and bioavailability with the aim to improve human health.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older

Exclusion Criteria:

* • Blood levels of HbA1c ≥ 6.5%, total cholesterol ≥ 240 mg/dL, LDL cholesterol ≥ 130 mg/dL, triglycerides ≥ 200 mg/dL

  * Are anemic (hemoglobin less than 13.5 g/dL in men and 12.0 g/dL in women)
  * Have an average blood pressure greater than or equal to 130/80 mmHg, or have diagnosed hypertension, hyperlipidemia, cardiovascular disease, diabetes, cancer, kidney, liver, gastrointestinal or pancreatic disease
  * Taking blood pressure-, lipid- or glucose-lowering, or hormone replacement medications
  * Are pregnant or are trying to become pregnant
  * Have a body mass index < 18.5 or > 30 kg/m2
  * >3 days/week vigorous exercise
  * Are not willing to maintain your normal eating/drinking and exercise habits over the duration of the study
  * History of smoking cigarettes in past 12 months
  * Binge and/or heavy drinker (>3 drinks on any given occasion and/or >7 drinks/week for women, and >4 drinks on any given occasion and/or >14 drinks/week for men)
  * Have allergies or contraindication to study treatments, procedures, or procedure supplies
  * Unable to attend study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Plasma polyphenol metabolites | Change from 0 hours (pre-treatment consumption) to 1 hour post-treatment consumption
  Plasma polyphenol metabolite analysis using mass spectrometry
Plasma polyphenol metabolites | Change from 0 hours (pre-treatment consumption) to 2 hours post-treatment consumption
  Plasma polyphenol metabolite analysis using mass spectrometry
Plasma polyphenol metabolites | Change from 0 hours (pre-treatment consumption) to 4 hours post-treatment consumption
  Plasma polyphenol metabolite analysis using mass spectrometry
Plasma polyphenol metabolites | Change from 0 hours (pre-treatment consumption) to 6 hours post-treatment consumption
  Plasma polyphenol metabolite analysis using mass spectrometry
Plasma polyphenol metabolites | Change from 0 hours (pre-treatment consumption) to 24 hours post-treatment consumption
  Plasma polyphenol metabolite analysis using mass spectrometry

SECONDARY OUTCOMES:
Urine polyphenol metabolites | 0 hours (pre-treatment consumption) and 24 hours post-treatment consumption
  Urine polyphenol metabolite analysis using mass spectrometry

OTHER OUTCOMES:
Gut microbial analysis | 0 hours (pre-treatment consumption) and 24 hours post-treatment consumption
  16S rRNA gene sequencing
Blood pressure | 0 hours (pre-treatment consumption) and 1, 2, 4, and 6 hours post-treatment consumption
  Brachial blood pressure parameters (systolic, diastolic, and pulse pressure)
Aortic pressure | 0 hours (pre-treatment consumption) and 1, 2, 4, and 6 hours post-treatment consumption
  Aortic pressure parameters (systolic pressure, aortic pressure, pulse pressure)
Augmentation index | 0 hours (pre-treatment consumption) and 1, 2, 4, and 6 hours post-treatment consumption
  Augmentation index measured via SphygmoCor Xcel
Glucose | 0 hours (pre-treatment consumption) and 1, 2, 4, 6, and 24 hours post-treatment consumption
  Blood glucose will be assessed using standard assays
Insulin | 0 hours (pre-treatment consumption) and 1, 2, 4, 6, and 24 hours post-treatment consumption
  Blood insulin will be assessed using standard assays
Nitric oxide metabolites | 0 hours (pre-treatment consumption) and 1, 2, 4, 6, and 24 hours post-treatment consumption
  Blood nitric oxide metabolites will be assessed using standard assays

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Johnson, PhD, RDN, Principal Investigator — Colorado State University, Department of Food Science and Human Nutrition; Charlene Van Buiten, PhD, Principal Investigator — Colorado State University, Department of Food Science and Human Nutrition
Locations (1):
- Food and Nutrition Clinical Research Laboratory - CSU Gifford Building, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chima B, Mathews P, Morgan S, Johnson SA, Van Buiten CB. Physicochemical Characterization of Interactions between Blueberry Polyphenols and Food Proteins from Dairy and Plant Sources. Foods. 2022 Sep 14;11(18):2846. doi: 10.3390/foods11182846. PMID 36140972